CLINICAL TRIAL: NCT04928196
Title: Evaluation of Retinal Microvasculature Before and After Silicone Oil Removal by Optical Coherence Tomography Angiography
Brief Title: Retinal Microvasculature Before and After Silicone Oil by OCTA
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Hebatalla Makled, Ophthalmology lecturer, Kasr El Aini Hospital
Other Study IDs: 6-1-2021-1
Record Dates: First submitted 2021-06-05; First posted 2021-06-16 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Retinal Vascular
Keywords: retinal microvasculature; microperimtry; OCTA; Silicone oil

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Microperimtery and optical coherence tomography angiography OCTA — observational: Investigations are done to assess the retinal microvasculature and function before and after silicone oil removal

SUMMARY:
Prospective study to assess the retinal microvasculature, optic nerve head vasculature and retinal sensitivity using OCTA and microperimetry before and after silicone oil removal.

DETAILED DESCRIPTION:
Prospective study to assess the retinal microvasculature, optic nerve head vasculature and retinal sensitivity using OCTA and microperimetry before and after silicone oil removal.

The study includes 30 patients with silicone oil tamponade will be evaluated before and after silicone oil removal

ELIGIBILITY:
Inclusion Criteria:

* 30 eyes of 30 patients with silicone oil tamponade will be evaluated before and after silicone oil removal

Exclusion Criteria:

* Proliferative diabetic retinopathy, recurrent detachment or macular hole
* Patients with chorioretinal degenerations involving the macula
* Secondary complications as cataract, silicone oil emulsification, or secondary glaucoma
* Media opacity hindering proper imaging

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Prospective observational case series of patients before and after silicone oil removal
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Macular and optic nerve head vascular density | one year
  Using OCTA to assess vascular density changes of the macula and optic nerve head before and after silicone oil removal
Retinal sensitivity by microperimetry | one year
  Using microperimetry to assess the retinal sensitivity changes before and after silicone oil removal

SECONDARY OUTCOMES:
Retinal vascular density and best corrected visual acuity | one year
  Correlate the change in the retinal vascular density with best corrected visual acuity
Optic nerve head vascular density and best corrected visual acuity | one year
  Correlate the change in the optic nerve head vascular density with best corrected visual acuity
Retinal sensitivity and best corrected visual acuity | one year
  Correlate the change in the retinal sensitivity with best corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Hebatalla S. Makled, MD, Principal Investigator — Kasr El Aini Hospital; Ghada A. Nassar, MD, Principal Investigator — Kasr El Aini Hospital; Maha M. Youssef, MD, Principal Investigator — Kasr El Aini Hospital; Lameece M. Hassan, MD, Principal Investigator — Kasr El Aini Hospital
Locations (1):
- Cairo University teaching hospital, Cairo, Egypt

REFERENCES:
- [Derived] Nassar GA, Makled HS, Youssef MM, Hassan LM. Functional and perfusion changes associated with silicone oil tamponade after macula-off rhegmatogenous retinal detachment surgery: an optical coherence tomography angiography/microperimetry study. Int Ophthalmol. 2024 Feb 22;44(1):107. doi: 10.1007/s10792-024-03037-5. PMID 38386180